CLINICAL TRIAL: NCT01422200
Title: Comparison of the Immunogenicity of Intramuscular Versus Subcutaneous Administration of Trivalent Inactivated Influenza Vaccine in Individuals With Neuromuscular Diseases
Brief Title: Flu Vaccine Study in Neuromuscular Patients 2011
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-2319
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Duchenne Muscular Dystrophy; Spinal Muscular Atrophy; Congenital Muscular Dystrophy
Keywords: DMD; SMA; CMD; flu vaccine
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant, care provider, and investigator are not masked. The outcomes assessor (personnel determining the HI titers) is masked.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous (Experimental): 0.5 mL of Fluzone (2011-2012 Northern Hemisphere formulation) influenza vaccine administered via subcutaneous route once
  Interventions: Biological: 2011-2012 seasonal flu vaccine Subcutaneous
- Intramuscular (Active Comparator): 0.5 mL of Fluzone (2011-2012 Northern Hemisphere formulation) influenza vaccine administered via intramuscular route once
  Interventions: Biological: 2011-2012 seasonal flu vaccine Intramuscular

INTERVENTIONS:
Biological: 2011-2012 seasonal flu vaccine Subcutaneous
  Other Names: fluzone
  Arms: Subcutaneous
Biological: 2011-2012 seasonal flu vaccine Intramuscular
  Other Names: fluzone
  Arms: Intramuscular

SUMMARY:
The purpose of the study is to compare the immune response of two different injection methods (Intramuscular V.S. Subcutaneous) of the 2011-2012 seasonal Influenza (Flu) vaccine among patients with neuromuscular conditions who have significant muscle degeneration. This research study hypothesizes that the subcutaneous route of vaccine administration, as compared to the intramuscular route, may confer at least comparable, or possibly better, immunogenicity. At least 30 individuals followed by the CCHMC Neuromuscular Comprehensive Care Center will be recruited to participate in this study lasting approximately one to two months with two clinic visits and one follow-up telephone call. Immunogenicity will be assessed by comparing hemagglutination inhibition (HI) antibody titers obtained pre- and post-vaccination.

DETAILED DESCRIPTION:
Individuals with neuromuscular diseases are more prone to influenza-related morbidity. Vaccination is the most effective measure to reduce the influenza disease burden. In the United States, the recommended route of administration for the inactivated influenza vaccine is intramuscular. In other countries, the subcutaneous, deep subcutaneous, and intramuscular routes are all considered acceptable for influenza vaccine administration. The United States CDC states that subcutaneous influenza vaccine doses, provided they are age-appropriate, may be counted as valid.

Those with neuromuscular diseases have muscle fibrosis that may potentially make intramuscular vaccines more effective. Those with Duchenne muscular dystrophy receive systemic corticosteroids to reduce inflammation. Corticosteroids may suppress antibody responses to vaccines. The goal of this research study is to evaluate the immunogenicity and safety of intramuscular and subcutaneous administration of inactivated influenza vaccine in individuals with neuromuscular diseases. This is a single site, open-label, randomized study. At the first visit, a blood sample was collected prior to vaccination. Each subject received either an intramuscular or subcutaneous vaccine administered in the anterolateral aspect of the thigh. Within 30 minutes of vaccination, subjects rated pain at the injection site using a numeric pain scale (0-10). Subjects and their caregivers were also asked to record local and systemic adverse events on diary sheets from day 0 to day 4 after vaccination. Subjects were instructed to notify the study staff by telephone should they develop any serious adverse reactions following vaccination. At a second study visit approximately 28 days later, a repeat blood sample was obtained. The blood samples obtained pre-vaccination and also at day 28 were tested for hemagglutination inhibition (HI) titers to the three influenza vaccine strains. rovider's office. The geometric mean titer ratios for each of the three vaccine strains were calculated as the ratios of postvaccination to prevaccination titers at geometric mean scale.

ELIGIBILITY:
Inclusion Criteria:

* Non-ambulatory;
* Quadriceps muscle strength of MRC (Medical Research Council Scale) grade 3 or below
* Any subject who is between 3 to 8 years of age must have received at least two doses of influenza vaccine last season or at least one dose tow or more years ago.

Exclusion Criteria:

* Subject must not have a history of severe reactions following previous immunization with influenza vaccine.
* Subject must not have previously received a 2011-2012 influenza vaccine.
* Subject must not have a history of Guillain-Barre syndrome.
* Subject must not have received a live viral vaccine (i.e., MMR, varicella) within 28 days prior to receipt of the study vaccine.
* Subject must not have any condition that the investigator believes would render vaccination unsafe or interfere with successful completion of the study.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Wong, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous; Intramuscular: 2011-2012 Northern Hemisphere formulation trivalent inactivated influenza vaccine
Period: Overall Study
Arm/Group | Subcutaneous | Intramuscular
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subcutaneous; Intramuscular: 2011-2012 Northern Hemisphere formulation inactivated influenza vaccine
- Total: Total of all reporting groups
Arm/Group | Subcutaneous | Intramuscular | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] — 10-28 years range
  years | 18.20 (4.88) | 19.37 (4.23) | 18.78 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer Ratio for Each Vaccine Strain
Description: Serum HI antibody titers for each vaccine strain immediately prior to study vaccine receipt and 21-28 days after study vaccine receipt
Time Frame: immediately before vaccination and 21-28 days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer ratio
Groups:
- Subcutaneous: Subjects receiving 2011-2012 Northern Hemisphere trivalent inactivated influenza vaccine by subcutaneous route
- Intramuscular: Subjects receiving 2011-2012 Northern Hemisphere trivalent inactivated influenza vaccine
Arm/Group | Subcutaneous | Intramuscular
Number analyzed (Participants) | 11 | 11
geometric mean titer ratio
  HINI vaccine strain | 3.76 [2.31 to 6.11] | 3.53 [1.43 to 8.7]
  H3N2 vaccine strain | 2 [1.49 to 2.68] | 1.46 [0.94 to 2.25]
  B vaccine strain | 1.76 [1.24 to 2.5] | 2 [1.11 to 3.6]
Statistical Analysis 1: Comparison: Subcutaneous vs Intramuscular; Test type: Other; p < .05, t-test, 2 sided

2. Other Pre Specified Outcome: Safety: Summary of Local and Systemic Reactogenicity Symptoms
Description: For the 4 days following receipt of study vaccine (days 0 to 4), the following local reactions will be assessed: pain, redness, and swelling. The following systemic reactions will also be assessed: body ache, weakness, irritability, headache, and cough.
Time Frame: 4 days following receipt of study vaccine
Population: Subjects who completed the diary sheets
Measure: Count of Participants; unit: Participants
Groups:
- Subcutaneous: 0.5 mL of Fluzone (2011-2012 Northern Hemisphere formulation) influenza vaccine administered via subcutaneous route once
  2011-2012 seasonal flu vaccine: Subcutaneous flu vaccine
- Intramuscular: 0.5 mL of Fluzone (2011-2012 Northern Hemisphere formulation) influenza vaccine administered via intramuscular route once
  2011-2012 seasonal flu vaccine: Intramuscular flu vaccine
Arm/Group | Subcutaneous | Intramuscular
Number analyzed (Participants) | 8 | 10
Participants
  Pain | 4 | 5
  Redness | 1 | 1
  Swelling | 2 | 1
  Body ache | 0 | 1
  Weakness | 0 | 1
  Irritabiltity | 0 | 1
  Headache | 1 | 0
  Cough | 0 | 1

ADVERSE EVENTS:
Time Frame: Local and systemic adverse events were collected on diary sheets from day 0 to day 4 after vaccination. Serious adverse events were collected through the final study visit, about 28 days.
Description: Within 30 minutes of vaccination, subjects rated the painfulness using a picture or numeric pain scale. Subjects and their caregivers were also asked to record local and systemic adverse events on diary sheets from day 0 to day 4 after vaccination. A mild symptom is one which is easily tolerated, a moderate symptom causes interference with usual daily activities, and a severe symptom results in the inability to perform daily activities.
Groups:
- Intramuscular: 2011-2012 Northern Hemisphere formulation trivalent inactivated influenza vaccine administered once intramuscularly
- Subcutaneous: 2011-2012 Northern Hemisphere formulation trivalent inactivated influenza vaccine administered once via subcutaneous route
Arm/Group | Intramuscular | Subcutaneous
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intramuscular (N=11) | Subcutaneous (N=11)
Paine/tenderness (Skin and subcutaneous tissue disorders) | 5 | 4
Redness (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling (Skin and subcutaneous tissue disorders) | 1 | 2
Body Ache (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Irritability (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small sample size as a pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes